CLINICAL TRIAL: NCT00097565
Title: The National Lymphocare Study: An Observational Study of Treatment, Outcomes, and Prognosis in Patients With Follicular Non-Hodgkin's Lymphoma
Brief Title: An Observational Study of Treatment, Outcomes, and Prognosis in Patients With Follicular Non-Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: U2963n
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Lymphoma, Non Hodgkin
Keywords: Follicular Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This is a prospective, observational, longitudinal, multicenter study of patients with newly diagnosed follicular Non Hodgkin's Lymphoma (NHL) designed to delineate differences in clinical outcome by comparing the effectiveness and safety of common treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (unless the Institutional Review Board [IRB] has granted a waiver of consent)
* Signed Authorization for the Use and Disclosure of Health Information document
* Age ≥18 years
* Histologic documentation of follicular NHL, according to Revised European-American Lymphoma (REAL) classification system, as assessed by the local pathologist and treating physician
* Initial diagnosis of follicular B-cell NHL within 6 months prior to enrollment
* Availability of cancer-specific historical data points in the patient's medical records

Exclusion Criteria:

* Other indolent or histologic NHL subtypes
* Diagnosis of lymphoma > 6 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with follicular NHL will be recruited from participating managed care organizations, community physicians or practices, and academic centers throughout the United States.
Sampling Method: Non-Probability Sample
Enrollment: 2740 (Actual)
Dates: Start 2004-03 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cinical Trials, Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Nastoupil LJ, Sinha R, Byrtek M, Ziemiecki R, Zhou X, Taylor M, Friedberg JW, Link BK, Cerhan JR, Dawson K, Flowers CR. Outcomes following watchful waiting for stage II-IV follicular lymphoma patients in the modern era. Br J Haematol. 2016 Mar;172(5):724-34. doi: 10.1111/bjh.13895. Epub 2016 Jan 5. PMID 26729445
- [Derived] Wagner-Johnston ND, Link BK, Byrtek M, Dawson KL, Hainsworth J, Flowers CR, Friedberg JW, Bartlett NL. Outcomes of transformed follicular lymphoma in the modern era: a report from the National LymphoCare Study (NLCS). Blood. 2015 Aug 13;126(7):851-7. doi: 10.1182/blood-2015-01-621375. Epub 2015 Jun 23. PMID 26105149